CLINICAL TRIAL: NCT04900129
Title: Inhalation of Vapor With Medication (Diclofenac Sodium, Menthol, Methyl Salicylate and N-Acetyl Cysteine) Reduces Oxygen Need and Hospital Stay in COVID-19 Patients - A Case Control Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sher-E-Bangla Medical College (Other)
Responsible Party: Principal Investigator, Harendra Nath Sarker, Professor, Sher-E-Bangla Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SBMC|Barisal|2020|1896
Record Dates: First submitted 2021-05-18; First posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Covid19
Keywords: Vapor; RT-PCR; Oxygen Saturation
MeSH Terms: conditions — COVID-19 | interventions — Menthol; methyl salicylate

STUDY DESIGN:
Intervention Model Description: Methods: Case control study Population: Adult patients with RT-PCR +ve mild to moderate COVID 19. Severe and critical disease patients had been excluded from the study.
  Duration: One month Study Place: Corona unit, Sher-E-Bangla Medical College Hospital, Barishal. Sample Size: Total 43 patients (N). Among them study group (SG) had 27 respondents and control group (CG) had 16 respondents Materials: Suitable vapor producing electric teapot, medicine, pulse oximeter and a structured questionnaire
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group (Experimental): This group inhaled vapor containing Menthol 0.02%, Methyl salicylate 0.05%, N- Acetyl cysteine 1.2 gm%, and Diclofenac sodium 1gm% twice daily in addition to conventional treatment. That is, 100 gram of emulsion contain diclofenac sodium 1 gram, N-acetyl cysteine 1.2 gm, menthol 20 mg, and methyl salicylic acid 50 mg. These drugs have no systemic and local side effects in these small doses, though it may cause slight eye irritation.
  Interventions: Combination Product: Menthol 0.02%, Methyl salicylate 0.05%, N- Acetyl cysteine 1.2 gm%, and Diclofenac sodium 1gm%
- Control Group (No Intervention): This group inhaled plain aquatic vapor in addition to conventional treatment.

INTERVENTIONS:
Combination Product: Menthol 0.02%, Methyl salicylate 0.05%, N- Acetyl cysteine 1.2 gm%, and Diclofenac sodium 1gm% — inhaled vapor containing Menthol 0.02%, Methyl salicylate 0.05%, N- Acetyl cysteine 1.2 gm%, and Diclofenac sodium 1gm% twice daily in addition to conventional treatment. That is, 100 gram of emulsion contain diclofenac sodium 1 gram, N-acetyl cysteine 1.2 gm, menthol 20 mg, and methyl salicylic acid 50 mg.
  Arms: Study Group

SUMMARY:
Background: In the midst of the devastating COVID pandemic where there is no specific and effective treatment, traditional therapy may help to ease the patient's suffering. Inhalation of vapor (VP) is an essential home remedy for stuffy, running nose in common cold, influenza and sinusitis. Steam inhalation is helpful in destroying the capsid of the SARS-CoV-2 envelope and preventing infection. Vapor with diclofenac sodium, menthol, methyl salicylate and N-acetyl cysteine may augment this effect. Objective: To evaluate the effect of inhalation of vapor with medication and to compare with inhalation of vapor without medication. Methods and Materials: A case control study taken place in Corona unit, Sher-E-Bangla Medical College Hospital, Barishal. 43 patients with mild to moderate COVID-19 were participated in this study. All are RT-PCR positive cases. Among them 16 patients were in control group and 27 in study group. In study group they were given vapor with Diclofenac Sodium, Menthol, Methyl Salicylate and N-Acetyl Cysteine and control group they were given normal steam/aquatic vapor two times in a day.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be COVID 19 positive and having a lack of oxygen saturation.

Exclusion Criteria:

* All the patients who do not covid infected.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Inhalation of Vapor with Medication (Diclofenac Sodium, Menthol, Methyl Salicylate and N-Acetyl Cysteine) Reduces Oxygen Need and Hospital Stay in COVID-19 Patients - A Case Control Study | 4 weeks
  This study determined that after regular inhalation of vapor with above medication, oxygen saturation level increased in the study group 384.61% in the morning and 515.79% at night comparing the control group. Furthermore, patients of study group need to stay nearly 1 day less in hospital in comparison to control group.

CONTACTS AND LOCATIONS:
Locations (1):
- HN Sarker, Barishal, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang J, Hajizadeh N, Moore EE, McIntyre RC, Moore PK, Veress LA, Yaffe MB, Moore HB, Barrett CD. Tissue plasminogen activator (tPA) treatment for COVID-19 associated acute respiratory distress syndrome (ARDS): A case series. J Thromb Haemost. 2020 Jul;18(7):1752-1755. doi: 10.1111/jth.14828. Epub 2020 May 11. PMID 32267998
- [Background] Tang N, Li D, Wang X, Sun Z. Abnormal coagulation parameters are associated with poor prognosis in patients with novel coronavirus pneumonia. J Thromb Haemost. 2020 Apr;18(4):844-847. doi: 10.1111/jth.14768. Epub 2020 Mar 13. PMID 32073213
- [Background] Woyke S, Rauch S, Strohle M, Gatterer H. Modulation of Hb-O2 affinity to improve hypoxemia in COVID-19 patients. Clin Nutr. 2021 Jan;40(1):38-39. doi: 10.1016/j.clnu.2020.04.036. Epub 2020 Apr 28. PMID 32360083
- [Background] Poston JT, Patel BK, Davis AM. Management of Critically Ill Adults With COVID-19. JAMA. 2020 May 12;323(18):1839-1841. doi: 10.1001/jama.2020.4914. No abstract available. PMID 32215647
- [Background] Alhazzani W, Moller MH, Arabi YM, Loeb M, Gong MN, Fan E, Oczkowski S, Levy MM, Derde L, Dzierba A, Du B, Aboodi M, Wunsch H, Cecconi M, Koh Y, Chertow DS, Maitland K, Alshamsi F, Belley-Cote E, Greco M, Laundy M, Morgan JS, Kesecioglu J, McGeer A, Mermel L, Mammen MJ, Alexander PE, Arrington A, Centofanti JE, Citerio G, Baw B, Memish ZA, Hammond N, Hayden FG, Evans L, Rhodes A. Surviving Sepsis Campaign: guidelines on the management of critically ill adults with Coronavirus Disease 2019 (COVID-19). Intensive Care Med. 2020 May;46(5):854-887. doi: 10.1007/s00134-020-06022-5. Epub 2020 Mar 28. PMID 32222812
- [Background] Griffiths MJD, McAuley DF, Perkins GD, Barrett N, Blackwood B, Boyle A, Chee N, Connolly B, Dark P, Finney S, Salam A, Silversides J, Tarmey N, Wise MP, Baudouin SV. Guidelines on the management of acute respiratory distress syndrome. BMJ Open Respir Res. 2019 May 24;6(1):e000420. doi: 10.1136/bmjresp-2019-000420. eCollection 2019. PMID 31258917
- [Background] Mairbaurl H, Weber RE. Oxygen transport by hemoglobin. Compr Physiol. 2012 Apr;2(2):1463-89. doi: 10.1002/cphy.c080113. PMID 23798307
- [Background] Dempsey JA. With haemoglobin as with politics - should we shift right or left? J Physiol. 2020 Apr;598(8):1419-1420. doi: 10.1113/JP279555. Epub 2020 Mar 13. No abstract available. PMID 32052863
- [Background] Mairbaurl H. Red blood cell function in hypoxia at altitude and exercise. Int J Sports Med. 1994 Feb;15(2):51-63. doi: 10.1055/s-2007-1021020. PMID 8157369
- [Result] de Wit E, van Doremalen N, Falzarano D, Munster VJ. SARS and MERS: recent insights into emerging coronaviruses. Nat Rev Microbiol. 2016 Aug;14(8):523-34. doi: 10.1038/nrmicro.2016.81. Epub 2016 Jun 27. PMID 27344959

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-05-23): https://cdn.clinicaltrials.gov/large-docs/29/NCT04900129/SAP_000.pdf